CLINICAL TRIAL: NCT05565326
Title: Pilot Study on Response Assessment During MR-guided Radiation Therapy for Glioblastoma Multiforme
Brief Title: Response Assessment During MR-guided Radiation Therapy for Glioblastoma
Acronym: MARGA
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Michael Mayinger, MD, University of Zurich
Other Study IDs: 2021-D0066
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Low field (0.35 T) MR-images of the brain at a MRIdian® linac system — Low field (0.35 T) MR-images of the brain at a MRIdian® linac system using CE marked low-field MR coils as provided by the company will be taken for volunteers in phase I. In phase II and III, after therapy beginning those images will be taken once per week per subject using CE marked low-field MR coils as provided by the company. This is done over the entire course of radiotherapy, which takes between 3 and 6 weeks.

SUMMARY:
The study seeks to assess the response of glioblastoma multiforme to treatment using weekly low field (0.35 T) MR-images of the brain at a MRIdian® linac system during standard radiotherapy at the same system. A total of 20 patients in a single arm will be recruited for this investigation.

The imaging data will be used to evaluate the change in tumor volume over the course of the treatment and to perform radiomics in order to investigate the possibility of response prediction using these images.

In order to assure sufficient image quality, prior to the main investigation, a group of up to 20 volunteers has MR scans taken with identical sequences to the main study phase.

ELIGIBILITY:
Inclusion criteria patients:

Subjects fulfilling all of the following criteria are eligible for the study:

* Informed Consent as documented by signature according to Swiss law and ICH/GCP regulations before any trial specific procedures (Appendix I Informed Consent Form)
* Histologically confirmed diagnosis of GBM
* Indication for fractionated radiation therapy for GBM
* Age: ≥ 18 years old
* Gender: any
* Karnofsky performance status ≥60
* Patients who are willing and able to comply with scheduled visits, treatment, and other trial procedures

Exclusion criteria

* The presence of any one of the following criteria will lead to exclusion of the subject:
* Previous cranial radiation therapy
* Contraindications to MR examinations, e.g., non-compatible implantable device or metallic foreign bodies
* Inability to complete MR examination due to claustrophobic anxiety
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: Female subjects of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Female subjects who are surgically sterilized / hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, diabetes, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glioblastoma patients undergoing radio(chemo)therapy.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess target volume changes with MRI during fractionated MR-guided radiation therapy. | 6 Months

SECONDARY OUTCOMES:
Value of target changes with MRI during fractionated MR-guided radiation therapy | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No